CLINICAL TRIAL: NCT02806219
Title: Open-label, Single-center, Randomized, Parallel Group, Single-dose, Bioequivalence Study of Certolizumab Pegol 200 mg Solution Injected Either by a Prefilled Syringe (Reference) or by an E-Device (Test) in Healthy Subjects
Brief Title: Open-label, Bioequivalence Study of Certolizumab Pegol 200 mg Solution Injected Either by a Prefilled Syringe (Reference) or by an E-Device (Test) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RA0132
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Certolizumab pegol; Human Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Certolizumab Pegol injection by prefilled syringe (Active Comparator)
  Interventions: Device: Prefilled syringe (PFS)
- Certolizumab Pegol injection by e-Device (Experimental)
  Interventions: Device: e-Device

INTERVENTIONS:
Device: Prefilled syringe (PFS) — Active substance: Certolizumab Pegol Pharmaceutical form: Solution for injection Administration: By prefilled syringe (PFS)
  Arms: Certolizumab Pegol injection by prefilled syringe
Device: e-Device — Active substance: Certolizumab Pegol Pharmaceutical form: Solution for injection Administration: By e-Device
  Arms: Certolizumab Pegol injection by e-Device

SUMMARY:
This is a single center, open-label, Phase 1 bioequivalence (BE) study in healthy subjects designed to demonstrate the bioequivalence of a single dose of certolizumab pegol (CZP) 200mg when injected by means of a prefilled syringe (PFS, reference) or injected by means of a injection device (e-Device, test).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between 18 and 55 years of age at Screening.
* Subject is in good physical and mental health status determined on the basis of the medical history and a general clinical examination.
* Subject has no evidence of active or inactive Tuberculosis (TB).
* Female subjects of childbearing potential should have a negative pregnancy test at study entry and should be using a medically accepted method of contraception during the entire duration of the study and for 10 weeks after the final dose of CZP.

Female subjects who are postmenopausal for at least 2 years and have a serum follicle stimulating hormone (FSH) level >40mIU/mL at the Screening Visit, or have undergone a hysterectomy, bilateral tubal ligation, and/or bilateral ovariectomy, or have a congenital sterility are considered not of childbearing potential.

Exclusion Criteria:

* Subject receiving any live (includes attenuated) vaccination or immunoglobulins within 56 days preceding the CZP injection.
* Subject has taken any drugs (including over-the-counter medications) within 56 days preceding the CZP injection (with the exception of those noted in Section 7.8.1.).
* Subject is known to be intolerant to pegol.
* Subject has previously received CZP.
* Subject has received TNFα-inhibitors within 12 months or other biologic within 6 months before randomization into the study.
* Subject has an active or chronic/latent infection including TB, hepatitis C virus (HCV), hepatitis B core antigen (HBc), or human immunodeficiency virus (HIV).-- Subject has symptomatic herpes zoster infection (shingles) within 6 months prior to Screening.
* Subject has chronic, serious, opportunistic recurring infection or condition within 6 months prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.
Area under the CZP plasma concentration-time curve from time 0 to infinity (AUC) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.
Area under the CZP plasma concentration-time curve from time 0 to last observed quantifiable concentration (AUC(0-t)) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.

SECONDARY OUTCOMES:
Time of observed Cmax (tmax) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.
Terminal elimination half-life (t1/2) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.
Apparent total body clearance (CL/F) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.
Apparent volume of distribution (Vz/F) | Predose on Day 1 and at 12 hours postdose, and on days 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 42, 56, 70.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB Pharma
Locations (1):
- Ra0132 001, Baltimore, Maryland, United States